CLINICAL TRIAL: NCT01211275
Title: A Randomized Phase I/II Study of Standard Chemotherapy (Cisplatin and Pemetrexed) With or Without Axitinib in Patients With Malignant Mesothelioma: Interim Biopsy Analysis to Determine Efficacy
Brief Title: Standard Chemotherapy With of Without Axitinib in Malignant Mesothelioma
Acronym: N08CPA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL25655.031.08
Record Dates: First submitted 2010-09-27; First posted 2010-09-29 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: mesothelioma; chemotherapy; translational research; axitinib
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma | interventions — Axitinib; Cisplatin; Pemetrexed; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- arm 2 (Experimental): axitinib + cisplatin + premetrexed
  Interventions: Biological: axitinib
- arm 1 (Active Comparator): cisplatin + premetrexed
  Interventions: Drug: chemotherapy

INTERVENTIONS:
Biological: axitinib — axitinib: 5 mg BID, day 2 until day 21 of each cycle; cisplatin: 75 mg/m2 day 1, every 3 weeks; pemetrexed: 500 mg/m2 day 1, every 3 weeks.
  Other Names: cisplatin; alimta
  Arms: arm 2
Drug: chemotherapy — cisplatin: 75 mg/m2 day 1, every 3 weeks; pemetrexed: 500 mg/m2 day 1, every 3 weeks.
  Other Names: cisplatin; alimta
  Arms: arm 1

SUMMARY:
The purpose of this study is to investigate the effects of axitinib, a potent angiogenesis inhibitor, on tissue and clinical outcome in combination with chemotherapy given to patients with mesothelioma

DETAILED DESCRIPTION:
To determine the effects of the addition of axitinib to standard chemotherapy on tissue samples with respect to micro-vessel density (MVD): expression of VEGF-Receptor; PDGF receptor expression; extent of necrosis and apoptosis.

To determine the safety of the addition of axitinib (to a maximum of the recommended dose of maximally 2 x 10 mg per day) to the standard treatment with cisplatin and pemetrexed.

To determine the feasibility of performing a (second) thoracoscopy after 10 weeks of the combination treatment with cisplatin, pemetrexed and axitinib.

Serum samples will be collected and tested for inhibiting effects in a tube formation and spheroid sprouting assay.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically diagnosed malignant mesothelioma
* age > 18 years
* Medically suitable for limited surgical intervention (pleural biopsies or limited pleurectomy)
* Measurable or evaluable disease is not required
* Ability to understand the study and give signed informed consent including the approval to accept a second thoracoscopic or surgical treatment after the third course
* No previous chemotherapy
* Radiotherapy is allowed when this is given for palliation, the interval is > 4 weeks, not more than 1/3 of the bone marrow capacity or all tumor is within the irradiation field.
* WHO performance status =< 2
* Adequate organ function as evidenced by the following peripheral blood counts or serum chemistries at study entry:

Hematology:

* ANC=>1.5 x 109/L,
* Platelets=>150 x 109/L,
* Hemoglobin => 6,0 mmol/l

Chemistry:

* total serum bilirubin < UNL;
* AST and ALT= < 2.5xUNL,
* AP < 5xUNL (unless bone metastases are present in the absence or any liver disease)
* Serum creatinine =< 2xUNL

Exclusion Criteria:

* Active uncontrolled infection, severe cardiac dysfunction or uncorrectable bleeding tendency
* Previous successful pleurodesis
* Uncontrolled hypertension
* Symptomatic peripheral neuropathy => grade 2 according to NCIC CTC,version 3.0
* Presence of symptomatic CNS metastases
* Unstable peptic ulcer, unstable diabetes mellitus or other serious disabling condition
* Concomitant administration to any other experimental drugs under investigation
* Impaired renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-05-22 (Actual); Primary Completion 2012-11-13 (Actual); Study Completion 2013-05-06 (Actual)

PRIMARY OUTCOMES:
To test the impact of the addition of axitinib to standaard chemotherapy treatment on histology samples | micro-vessel density;expression of VEGF and PDGF receptor; extent of necrosis and apoptosis
  To determine the effects of the addition of axitinib to standard chemotherapy on tissue samples with respect to micro-vessel density (MVD); expression of VEGF-Receptor; PDGF receptor expression; extent of necrosis and apoptosis

SECONDARY OUTCOMES:
the side effects of the standard chemotherapy and the additional risks related to axitinib use | AE;SAE;SUSAR
  hypertension, fatigue, abdominal discomfort

CONTACTS AND LOCATIONS:
Overall Officials: P Baas, Dr., Principal Investigator — NKI-AvL
Locations (1):
- Antoni van Leeuwenhoekziekenhuis (NKI-AVL), Amsterdam, North Holland, Netherlands